CLINICAL TRIAL: NCT03703115
Title: The Effect of Fasting on ICSI Outcomes in Patients With Polycystic Ovary Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no commitment from the patient to maintain fasting in both the control and case groups
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdel-Maguid Ramzy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 88766603
Record Dates: First submitted 2018-09-29; First posted 2018-10-11 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2021-01

CONDITIONS: Infertility; Polycystic Ovary Syndrome
Keywords: ICSI; Polycystic ovary syndrome; Infertility; Fasting
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome; Fasting | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (Active Comparator): Patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet with 2-3 litres of water and non calorie fluids allover the day.
  Interventions: Behavioral: Fasting
- Nonfasting (No Intervention): Patients will have usual balanced diet as 3 meals and 2 snacks all over the day. Both groups should take adequate water and non calorie beverages intake daily ( 2-3 liters daily)

INTERVENTIONS:
Behavioral: Fasting — No food for 14 -16 hours with water intake and non caloric beverages then eating balanced meals over 8 to 10 hours
  Other Names: Periodic fasting
  Arms: Fasting

SUMMARY:
Design and protocol of PCO fasting research:

This study is a pilot prospective, single-blinded (to the health assessor), randomized controlled trial conducted at the In Vitro Fertilization ( IVF) center of the Department of Obstetrics & Gynecology, Kasr El-Ainy Hospital, Cairo University, Egypt, from October 2018 to September 2019, to determine the clinical effect of fasting on ICSI outcomes in PCOS patients. Ethical committee approval was obtained. The study will include 100 infertile patients with PCOS diagnosed according to Rotterdam criteria of PCOS and who are candidates for ICSI cycle. Women with diabetes, thyroid disorder or other endocrine dysfunctions, uterine abnormalities were excluded.

All patients are informed about the study and consent is given by those who accept to participate.

Careful history taking include infertility type, duration , cause, obstetric history, medical and surgical history and demographic distribution is taken. Full physical examination and 2 dimensional (2D) transvaginal sonography (TVS) are done on day 2 to 5 of menses to assess antral follicle count, uterus and adnexa . Body mass index (BMI) and waist/hip ratio (WHR) are calculated, Blood samples are taken for Fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA index), lipid profile and hormonal profile are done.

All 100 participants will be randomized withdrawing closed envelopes for each patient into group A and group B .

Group (A): patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. Group (B): no fasting, patients will have usual balanced diet as 3 meals and 2 snacks all over the day. Both groups should take adequate water and non calorie beverages intake daily (2-3 liters) Subjects are instructed to wait for spontaneous menses, or to be prescribed progestins orally (as Norethisterone 5mg) twice daily for 21 days starting from the fifth day of menses. Patients should continue taking oral metformin 500-1000 mg daily, until confirmation of pregnancy.

The next visit is scheduled on day 2 of next cycle when transvaginal ultrasound is done to confirm that endometrial thickness <5mm, no ovarian cyst by ultrasound. Body mass index (BMI) and waist/hip ratio (WHR) are calculated. Blood samples are taken for Fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG), Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2),and then antagonist protocol is followed. Gonadotropins as Intramuscular (I.M.) injections of 150-300 (International units) I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). and Urofollitropin or highly purified human follicle stimulating hormone(Fostimon®, 75 I.U. /vial, IBSA) are give in a ratio of 1:1.The dose is adjusted according to the age, BMI, Antral follicle count (AFC), serum levels of AMH, FSH and ovarian response.

Fixed antagonist protocol is given and follow up until embryo transfer(ET). Quantitative ß- HCG in serum after is done after 14 days of embryo transfer.TVS is performed to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile and other ICSI outcomes.

DETAILED DESCRIPTION:
Design and protocol of PCO fasting research:

This study is a pilot prospective, single-blinded (to the health assessor), randomized controlled trial conducted at the In Vitro Fertilization ( IVF) center of the Department of Obstetrics & Gynecology, Kasr El-Ainy Hospital, Cairo University, Egypt, from October 2018 to September 2019, to determine the clinical effect of fasting on ICSI outcomes in PCOS patients. Ethical committee approval was obtained. The study will include 100 infertile patients with PCOS diagnosed according to Rotterdam criteria of PCOS and who are candidates for ICSI cycle. Women with diabetes, thyroid disorder or other endocrine dysfunctions, uterine abnormalities were excluded.

All patients are informed about the study and consent is given by those who accept to participate.

Careful history taking include infertility type, duration , cause, obstetric history, medical and surgical history and demographic distribution is taken. Full physical examination and 2 dimensional (2D) transvaginal sonography (TVS) are done on day 2 to 5 of menses to assess antral follicle count, uterus and adnexa . Body mass index (BMI) and waist/hip ratio (WHR) are calculated, Blood samples are taken for Fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA index), lipid profile ( Triglycerides, total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG), Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2) All 100 participants will be randomized withdrawing closed envelopes for each patient into group A and group B .

Group (A): patients will have periodic fasting for 4 weeks prior to the treatment cycle. The fasting method involves daily fasts of 14-16hours and restrict eating to an 8-10 hour "eating window" as 2-3 or more meals of balanced diet. Group (B): no fasting, patients will have usual balanced diet as 3 meals and 2 snacks all over the day. Both groups should take adequate water and non calorie beverages intake daily (2-3 liters) Subjects are instructed to wait for spontaneous menses, or to be prescribed progestins orally (as Norethisterone 5mg) twice daily for 21 days starting from the fifth day of menses. Patients should continue taking oral metformin 500-1000 mg daily, until confirmation of pregnancy.

The next visit is scheduled on day 2 of next cycle when transvaginal ultrasound is done to confirm that endometrial thickness <5mm, no ovarian cyst by ultrasound. Body mass index (BMI) and waist/hip ratio (WHR) are calculated. Blood samples are taken for Fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG), Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2),and then antagonist protocol is followed. Gonadotropins as Intramuscular (I.M.) injections of 150-300 (International units) I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). and Urofollitropin or highly purified human follicle stimulating hormone(Fostimon®, 75 I.U. /vial, IBSA) are give in a ratio of 1:1.The dose is adjusted according to the age, BMI, Antral follicle count (AFC), serum levels of AMH, FSH and ovarian response.

On the sixth day of stimulation , a visit is scheduled to assess the ovarian response ( folliculometry) by TVS. Gonadotrophin releasing hormone antagonist (GnRH antagonist) which is Cetrorelix 0.25mg ( Cetrotide®, 0.25 mg/ vial, Merck Serono, is filled and mixed with diluent from a prefilled syringe with a 20 gauge needle) is given subcutaneously (S.C.) by 27-gauge needle starting from the 6th day of stimulation (fixed antagonist protocol).

Next visits are every other day for follow up using the TVS. The trigger by Human Chorionic Gonadotrophin (HCG)10000 I.U., I.M. ( Pregnyl, Organon) is given when at least 3 follicles reach 18mm in mean diameter or more and E2 level is less than 2500 pg/ml. Ovum retrieval is done 34 hours after HCG injection and embryo transfer using Wallace catheter on day 2 to 3. Luteal support includes natural Progesterone 400 mg 1x2 as rectal suppository, Folic acid 0.5 mg orally once daily, Amoxicillin-Clavulanic Acid 1gm 1x2x7 orally, Progesterone 100 I.M. injections daily for 10 days, Acetylsalicylic Acid (75 mg) orally once daily, metformin 500-1000 mg orally daily .

Quantitative ß- HCG in serum after is done after 14 days of embryo transfer.TVS is performed to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG)u, Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2, Days of stimulation , dose of gonadotrophins, number of M II oocytes retrieved, number of grade1and 2 embryos, number of frozen embryos, freeze all cycles, Ovarian Hyperstimulation syndrome (OHSS), Chemical pregnancy rate, clinical pregnancy, twins, abortion, ectopic pregnancy, preterm labour, live birth rate

ELIGIBILITY:
Inclusion Criteria:

* infertile patients with polycystic ovary syndrome diagnosed according to the Rotterdam criteria scheduled for ICSI

Exclusion Criteria:

* women with diabetes, thyroid disorders and other endocrinologic disorders
* women with uterine abnormalities

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical pregnancy | 10 weeks
  detection of gestationalsac, embryonal pole and fetal pulsations by ultrasonography

SECONDARY OUTCOMES:
Body mass index | 4 weeks of fasting
  The weight in kilograms divided by the squared height in meters
Waist/ hip ratio | 4 weeks of fasting
  The ratio of waist circumference in centimeters to the hip circumference in centimeters
Concentration of fasting insulin | 4 weeks of fasting
  Insulin level in serum after fasting for 8 hours measured as mIU/ml
Concentration of free testosterone | 4 weeks of fasting
  Free testosterone level in serum measured as ng/dL
Number of days of stimulation with gonadotrophins | 6 weeks
  Days of stimulation with gonadotrophins
Number of ampoules of gonadotrophins | 6 weeks
  total number of ampoules of gonadotrophins
Number of M II oocytes retrieved | Average 6 weeks
  Number of M II oocytes retrieved
Number of grade1 and 2 embryos | 6-7 weeks
  Number of grade1 and 2 embryos
Number of frozen embryos | 6 to 7 weeks
  Number of frozen embryos
Number of freeze all cycles | 6 to 7 weeks
  total number of freeze all cycles
Number of cases with Ovarian Hyperstimulation Syndrome | 6 to 8 weeks
  number of cases diagnosed with Ovarian Hyperstimulation Syndrome
Rate of chemical pregnancy | 10weeks
  number of cases with positive pregnancy test with no clinical pregnancy
Rate of twin pregnancy | 10 weeks
  presence of two gestational sacs detected by ultrasonography
Rate of ectopic pregnancy | 10 weeks
  the presence of gestational sac outside the uterine cavity detected by ultrasound
Rate of Abortion | 10-24 weeks
  the number of abortions clinically diagnosed per cycle
Rate of preterm labour | After 24 weeks of start of study
  labour after 20 weeks of gestation and before completed 37 weeks of gestation
Rate of live birth | After40 weeks of start of study
  Live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Abdelmaguid Ramzy, Principal Investigator — Cairo University
Locations (1):
- KasrELAiniH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No